CLINICAL TRIAL: NCT02008240
Title: Salpingectomy Versus Aspiration of Hydrosalpingeal Fluid Prior to IVF-ET.A Randomized Controlled Trial
Brief Title: Salpingectomy Versus Aspiration of Hydrosalpingeal Fluid Prior to IVF-ET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Prof .Usama M.Fouda, M.D , PhD, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hydrosalpinx2
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Infertility
Keywords: Infertility; Hydrosalpinx; IVF-ET; Salpingectomy
MeSH Terms: conditions — Infertility | interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Needle aspiration of hydrosalpinx (Experimental): Aspiration of hydrosalpingeal fluid under ultrasound guidance
  Interventions: Procedure: Needle aspiration of hydrosalpinx
- salpingectomy (Active Comparator): Surgical removal of hydrosalpinx
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Needle aspiration of hydrosalpinx — Under deep sedation, the retrieval of oocytes is done and then an aspiration needle is inserted into the hydrosalpinx under ultrasonographic guidance and suction is applied to aspirate the hydrosalpingeal fluid completely . If there are bilateral hydrosalpinges, the process is repeated on the opposite side.
  Other Names: ultrasound guidance aspiration of hydrosalpingeal fluid
  Arms: Needle aspiration of hydrosalpinx
Procedure: Salpingectomy — laparoscopic surgical removal of affected tube is done with bipolar electrocoagulation for hemostasis. The mesosalpinx is coagulated as close a possible to the fallopian tube to avoid any compromise in the ovarian blood supply . In cases with marked adhesion, proximal ligation and a distal fenestration is done .
  Other Names: surgical removal of hydrosalpinx
  Arms: salpingectomy

SUMMARY:
The aim of this randomized controlled trial is to compare the efficacy of ultrasound guided aspiration of hydrosalpingeal fluid with salpingectomy in the management patients with ultrasound visible hydrosalpinges undergoing IVF-ET.

DETAILED DESCRIPTION:
The adverse impact of hydrosalpinx on in vitro fertilisation embryo transfer (IVF-ET) outcomes has been confirmed by several retrospective and prospective studies .

Cochrane review of prospective randomised trials of laparoscopic salpingectomy confirmed the beneficial effect of laparoscopic salpingectomy on IVF-ET outcomes in patients with hydrosalpinges.

Surgery is not usually safe especially in patients with extensive adhesions, morbid obesity or previous multiple laparotomies. Furthermore, many infertile couples refuse to undergo bilateral salpingectomy or proximal tubal occlusion because these procedures remove any hope of spontaneous pregnancy. Other less invasive options for patients with hydrosalpinges as ultrasound-guided aspiration of hydrosalpingeal fluid, antibiotics (alone or combined with aspiration) and hysteroscopic occlusion of fallopian tube were studied in order to find an alternative to salpingectomy . Although these methods are simple and getting popular, current data are inadequate to recommend these treatment options instead of salpingectomy because most of the supporting evidences for these methods come from small retrospective studies.

A recent randomized controlled trial revealed that the aspiration of hydrosalpingeal fluid at the time of oocyte retrieval was associated with improved implantation rate and pregnancy rates.

The aim of this randomized controlled trial is to compare the efficacy of ultrasound guided aspiration of hydrosalpingeal fluid with salpingectomy in the management patients with ultrasound visible hydrosalpinges undergoing IVF-ET

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral hydrosalpinges visible by ultrasound
* Age between 18 - 37 years
* Period of infertility > 1 year
* Body mass index between 19-29
* Normal basal luteinizing hormone (LH), follicle stimulating hormone (FSH) and prolactin concentrations.
* Normal recent semen analysis (according to World Health Organization criteria).

Exclusion Criteria:

* Uterine fibroid requiring surgical removal.
* Endometriosis.
* Male factor of infertility requiring ICSI, Previous IVF cycles.
* History of recurrent miscarriage.
* Endocrinologic disorders.
* Presence of systemic disease contraindicating pregnancy.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The Number of Participants Who Achieved Clinical Pregnancy in a Transfer Cycle | 5 weeks after embryo transfer

SECONDARY OUTCOMES:
The Number of Participants Who Achieved Ongoing Pregnancy in a Transfer Cycle . | 18 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Usama M. Fouda, M.D, PhD, Study Chair — Assistant professor of Obstetrics and Gynecology , Faculty of medicine ,Cairo university , and scientific director of assisted conception unit, Aljazeera (Al Gazeera) hospital.; Ahmed M. Sayed, M.D, PhD, Study Director — Assistant professor of Obstetrics and Gynecology , Faculty of medicine ,Cairo university, and clinical director of assisted conception unit, Aljazeera (Al Gazeera) hospital
Locations (1):
- Aljazeera (Al Gazeera) hospital, Giza, Giza Governorate, Egypt

REFERENCES:
- [Background] Fouda UM, Sayed AM. Effect of ultrasound-guided aspiration of hydrosalpingeal fluid during oocyte retrieval on the outcomes of in vitro fertilisation-embryo transfer: a randomised controlled trial (NCT01040351). Gynecol Endocrinol. 2011 Aug;27(8):562-7. doi: 10.3109/09513590.2010.507290. Epub 2010 Jul 30. PMID 20672903
- [Background] Strandell A, Lindhard A, Waldenstrom U, Thorburn J, Janson PO, Hamberger L. Hydrosalpinx and IVF outcome: a prospective, randomized multicentre trial in Scandinavia on salpingectomy prior to IVF. Hum Reprod. 1999 Nov;14(11):2762-9. doi: 10.1093/humrep/14.11.2762. PMID 10548619
- [Derived] Fouda UM, Sayed AM, Abdelmoty HI, Elsetohy KA. Ultrasound guided aspiration of hydrosalpinx fluid versus salpingectomy in the management of patients with ultrasound visible hydrosalpinx undergoing IVF-ET: a randomized controlled trial. BMC Womens Health. 2015;15:21. doi: 10.1186/s12905-015-0177-2. Epub 2015 Feb 27. PMID 25783650